CLINICAL TRIAL: NCT06453330
Title: A Randomised Control Clinical Trial Investigating the Effect of Horizontal-Platelet-Rich Fibrin (H-PRF) vs Standard Placement on Implant Stability and Marginal Bone Levels in Adults
Brief Title: A Randomised Control Clinical Trial Investigating the Effect of H-PRF on Implant Stability and Marginal Bone Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Rawan Kahatab, Postgraduate periodontology student, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3470
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Osseointegration Failure of Dental Implant

STUDY DESIGN:
Intervention Model Description: An intervention group receiving standard placement of single implants with H-PRF and a control group receiving standard placement of single implants without H-PRF
Masking Description: Due to the nature of having to draw blood from participants who will be receiving H-PRF, nobody can be masked/blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An intervention group receiving standard placement of single implants with H-PRF (Experimental): H-PRF preparation protocol involves taking a sample of venous blood from patients using a butterfly needle to collect up to 8-9ml tubes of blood. After the first tube is collected, it would immediately be placed in a horizontal centrifuge machine, balanced out with 3 tubes of water, to ensure the centrifuge is properly balanced. A set rpm and time will be chosen, and the centrifuge will run until the time is complete. The H-PRF clots would then be ready and taken out of the tubes to separate them from the red blood cells.
  Interventions: Biological: Horizontal platelet-rich fibrin (H-PRF)
- A control group receiving standard placement of single implants without H-PRF (No Intervention): this group will have standard implant placement without H-PRF

INTERVENTIONS:
Biological: Horizontal platelet-rich fibrin (H-PRF) — Most commercially available centrifuges used for PRF production are fixed-angle systems designed primarily for pelleting samples to the bottom of tubes and are not particularly efficient at separating the cell layers effectively. Research has demonstrated that PRF produced using horizontal centrifugation (H-PRF) can lead to a higher concentration of platelets and leukocytes compared to PRF produced from fixed-angle centrifugation (LPRF). The resulting PRF from horizontal centrifugation is termed 'horizontal platelet-rich fibrin' (H-PRF). The H-PRF clot will be produced using a Bio-PRF horizontal centrifuge machine. This machine is CE marked and regularly used in the Dublin Dental University Hospital.
  Arms: An intervention group receiving standard placement of single implants with H-PRF

SUMMARY:
This research will be a randomised controlled trial (RCT) investigating whether the use of Horizontal Platelet Rich Fibrin (H-PRF) increases implant stability compared to those implants placed without H-PRF, and therefore, contributes to the implant's overall success.

H-PRF is a second generation platelet concentrate that consists of a fibrin mesh containing cytokines and leukocytes. It has been shown to stimulate mesenchymal stem cells and osteoblasts that encourage bone formation as a result of the growth factors released from platelets, which should aid in osseointegration of implants. There is limited research that investigates the effects of H-PRF on implant stability. There is, however, some evidence that platelet-rich fibrin (PRF), which is produced in a fixed-angle centrifuge, increases implant stability and H-PRF is considered the evolution of PRF products.

This research would follow a H-PRF preparation protocol which involves taking a sample of venous blood from patients using a butterfly needle to collect up to 8-9ml tubes of blood. After the tube of blood is collected, it would immediately be placed in a horizontal centrifuge machine with 3 tubes of water to balance the centrifuge, and placed opposite each other. A set rpm and time will be chosen, and the centrifuge will run until the time is complete. The H-PRF clots would then be ready and taken out of the tubes to separate them from the red blood cells.

Following randomisation, implants will be placed in the upper or lower jaws of patients attending the Dublin Dental University Hospital using the standard implant protocol. Half of the implants will be coated with H-PRF, the other half (control group) would be placed without HPRF. Implant stability and marginal bone levels will be measured at three different stages: 1) Initial implant placement, 2) Second stage surgery when the implant is uncovered after healing and integrated with the bone, 3) When the definitive crown or bridge is attached to the implant. Insertion torque at baseline will also be measured. The above results will be collected and assessed to determine the effects of H-PRF, if any, on implant stability and the preservation of bone levels around implants.

DETAILED DESCRIPTION:
This is a parallel arm, randomised control clinical Trial (RCT) on a cohort of Dublin Dental University Hospital patients who are having dental implants placed in the maxilla or mandible.

Study sample:

1. Subjects will be recruited from a population of patients who have been referred to Dublin University Dental Hospital from general practice or specialist practice for provision of implants
2. Subjects will be recruited from a population of patients who have been referred from another department within the Dublin Dental Hospital for provision of implants.

Enrolment and Consent:

Participants will be selected via two methods:

1. Subjects will be recruited from a population of patients who have been referred to Dublin University Dental Hospital from general practice or specialist practice for provision of implants.
2. Subjects will be recruited from a population of patients who have been referred from another department within the Dublin Dental University Hospital for provision of implants. Patients being referred for implants to the Dublin Dental University hospital initially attend a dental implant assessment appointment. If at that appointment they are deemed suitable to be enrolled in the study, a gatekeeper, Ms Niamh Leonard, will invite the patient to take part in the research study. (Please note that Ms Niamh Leonard is an experienced gatekeeper and an administrator in the Division of Restorative Dentistry and Periodontology in the Dublin Dental Hospital, but is not involved in study patient's care. She will only be involved in inviting patients to take part in the study). Patients will have an opportunity to discuss the study in detail and will be provided with a written copy of the Patient Information Leaflet (PIL) to take home. For any question that may arise regarding the research or the surgical procedure patients will be able to contact the co-investigator (Dr Rawan Kahatab) as the contact details appear on the information leaflet. Patients will be given time (at least 7 days) to consider their participation and can contact the gatekeeper if they opt to participate. Patients will sign a freely given informed consent form prior to their enrolment in the study.

If a single patient will be receiving more than one dental implants and there are numerous implant sites that qualify for entry into the research, only one of the implant sites will be randomly selected for the study. If a patient opts not to participate, it will not affect their care.

Randomisation:

At the time of surgery, each patient will select a numbered, sealed envelope with the treatment group allocation. Each envelope will correspond to a number on a computer-generated randomisation list created prior to enrolment of study participants. The operator will then use either the H-PRF or not use H-PRF when placing the implant depending on what was revealed when the envelope was opened. Neither the operator or the patient can be blinded to the arm chosen as blood sample will only be taken for the H-PRF group.

The blood sample collection and surgeries will be performed by Dr Rawan Kahatab.

H-PRF is used regularly in the DDUH and the clinical protocol will not deviate from standard procedures used at the hospital. H-PRF preparation protocol involves taking a sample of venous blood from patients using a butterfly needle to collect up to 8-9ml tubes of blood. After the first tube is collected, it would immediately be placed in a horizontal centrifuge machine, balanced out with 3 tubes of water, to ensure the centrifuge is properly balanced. A set rpm and time will be chosen, and the centrifuge will run until the time is complete. The H-PRF clots would then be ready and taken out of the tubes to separate them from the red blood cells. Peri-apical radiographs of the surgical site are taken pre-operatively, at implant placement and at implant restoration for all implants placed at the Dublin Dental University Hospital.

________________________________________________________________

Similar studies that have previously been carried out to assess the effect of PRF on implant stability have focused on PRF produced from fixed-angle systems as opposed to horizontal ones. However, they have followed a very similar design to our proposed design. For example, in a study by Tabrizi et al., (2017), a split-mouth randomised clinical trial was performed. Twenty patients with missing teeth in the molar region of the maxilla, requiring bilateral implants, were included. PRF was used on one side (group 1); no PRF was used on the other (group 2). Implant stability was assessed by resonance frequency analysis (RFA) at 2, 4, and 6 weeks after placement. At 2 weeks, the mean ISQ was 60.60 ± 3.42 in group 1 and 58.25 ± 3.64 in group 2; at 4 weeks it was 70.30 ± 3.36 in group 1 and 67.15 ± 4.33 in group 2; at 6 weeks it was 78.45 ± 3.36 in group 1 and 76.15 ± 2.94 in group 2. Significant differences in RFA were found between the groups at 2 weeks (P = 0.04), 4 weeks (P = 0.014), and 6 weeks (P = 0.027) after placement.

The study results suggest that the use of PRF may enhance the post-insertion stability of dental implants placed in the posterior maxilla during the healing period. In another study by Oncu et al., (2015), twenty healthy patients with adequate alveolar bone and two or more adjacent missing teeth extracted at least 6 months previously were included. A minimum of two tapered implants were placed in each patient. After surgical preparation of the implant sockets, PRF that had been prepared preoperatively was placed randomly into one of the sockets. Resonance frequency measurements were made after implant placement and at 1 week and 1 month postoperatively. Mean implant stability quotients (ISQs) of the PRF implants was 69.3 ± 10.5, and mean ISQs for the PRF- implants was 64.5 ± 12.2 at the end of the first week. The mean ISQs at 4 weeks postoperatively were 77.1 ± 7.1 for the PRF+ group and 70.5 ± 7.7 for the group without PRF. In this study, PRF application increased implant stability during the early healing period, as evidenced by higher ISQ values. Based on the results of these studies and the fact that H-PRF is an even more superior biomaterial than PRF, our study should achieve outcomes that are just as successful.

ELIGIBILITY:
Inclusion Criteria:

Patient Level

* Male or Female, 18 years old or over
* Capacity to provide informed consent
* Willing to comply with study appointment schedule and willing to maintain a diary of symptoms
* Planned for provision of dental implant(s) at Dublin Dental University Hospital Site Level
* Sufficient bone volume for implant placement without the need for bone graft/augmentation; alveolar ridge of minimum 6mm width for standard implants (implant diameter 4mm) and of minimum 7mm for wider implants (implant diameter 5mm)

Exclusion Criteria:

Patient Level

* Plaque score >20%
* Bleeding score >20%
* Tobacco smoking
* Uncontrolled systemic disease
* Use of systemic medications with an expected impact on bone healing (e.g. bisphosphonates)
* Pregnancy or lactation
* Lack capacity to give informed consent
* History of radiotherapy to the head and/or neck Site Level
* Insufficient bone volume for implant placement, requiring bone graft/augmentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Implant Stability Quotient (ISQ) using magnetic resonance frequency analysis (MRFA) | At implant placement, at 3 months and at 4-5 months (implant restoration)
  This is a measurement of the stability of the implant

SECONDARY OUTCOMES:
Secondary outcomes: Marginal bone levels | At implant placement, at 3 months and at 4-5 months (implant restoration)
  The level of bone around the implant
Rate of pain experienced based on a visual analog scale 1-10 | after local anaesthetic wears away, 24 hours after implant placement and 1 week after implant placement
  Rate of pain experienced using a survey that will be given to patients. They will be given a visual analog scale and asked to use that to rate their pain.
Number of participants with implant loss/fracture/infection | At any point from implant placement until 4-5 months afterwards
  Any implant failures/infections. This includes loss of implant, fracture of the implant or infection of the implant site.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ioannis Polyzois, Consultant, Principal Investigator — Dublin Dental University Hospital
Locations (1):
- Dublin Dental University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
It is unlikely that patient data (Identification and personal details) will be shared, only the outcome measurements and details of where the implant was placed.

REFERENCES:
- [Background] Tabrizi R, Arabion H, Karagah T. Does platelet-rich fibrin increase the stability of implants in the posterior of the maxilla? A split-mouth randomized clinical trial. Int J Oral Maxillofac Surg. 2018 May;47(5):672-675. doi: 10.1016/j.ijom.2017.07.025. Epub 2017 Dec 18. PMID 29269149
- [Background] Oncu E, Alaaddinoglu EE. The effect of platelet-rich fibrin on implant stability. Int J Oral Maxillofac Implants. 2015 May-Jun;30(3):578-82. doi: 10.11607/jomi.3897. PMID 26009908
- [Background] Miron RJ, Chai J, Zheng S, Feng M, Sculean A, Zhang Y. A novel method for evaluating and quantifying cell types in platelet rich fibrin and an introduction to horizontal centrifugation. J Biomed Mater Res A. 2019 Oct;107(10):2257-2271. doi: 10.1002/jbm.a.36734. Epub 2019 Jun 12. PMID 31148358
- [Background] Lucarelli E, Beccheroni A, Donati D, Sangiorgi L, Cenacchi A, Del Vento AM, Meotti C, Bertoja AZ, Giardino R, Fornasari PM, Mercuri M, Picci P. Platelet-derived growth factors enhance proliferation of human stromal stem cells. Biomaterials. 2003 Aug;24(18):3095-100. doi: 10.1016/s0142-9612(03)00114-5. PMID 12895582
- [Background] Uggeri J, Belletti S, Guizzardi S, Poli T, Cantarelli S, Scandroglio R, Gatti R. Dose-dependent effects of platelet gel releasate on activities of human osteoblasts. J Periodontol. 2007 Oct;78(10):1985-91. doi: 10.1902/jop.2007.070116. PMID 18062120
- [Background] Anitua EA. Enhancement of osseointegration by generating a dynamic implant surface. J Oral Implantol. 2006;32(2):72-6. doi: 10.1563/736.1. PMID 16704108
- [Background] Fujioka-Kobayashi M, Kono M, Katagiri H, Schaller B, Zhang Y, Sculean A, Miron RJ. Histological comparison of Platelet rich fibrin clots prepared by fixed-angle versus horizontal centrifugation. Platelets. 2021 Apr 3;32(3):413-419. doi: 10.1080/09537104.2020.1754382. Epub 2020 Apr 18. PMID 32306811